CLINICAL TRIAL: NCT05745584
Title: Effect of Mirabegron on Bladder Compliance ; a Prospective Paired Comparison of Mirabegron and Anticholinergics in Patients With Low Bladder Compliance
Brief Title: Effect of Mirabegron on Bladder Compliance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2015-0938
Record Dates: First submitted 2023-02-03; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Patients With Low Bladder Compliance of 20ml/H2O or Less Despite Taking Anticholinergics
Keywords: Mirabegron; Beta3-adrenoceptor agonist; Bladder compliance
MeSH Terms: interventions — mirabegron; Cholinergic Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): 8 weeks of mirabegron treatment==> 8 weeks of anticholinergics treatment
  Interventions: Drug: Mirabegron (beta3-adrenoceptor agonist), Anticholinergics

INTERVENTIONS:
Drug: Mirabegron (beta3-adrenoceptor agonist), Anticholinergics — Administration of Mirabegron (beta3-adrenoceptor agonist) for 8 weeks, and followed by subsequent administration of anticholinergics for 8 weeks

SUMMARY:
In many cases of neurogenic bladder patients, bladder compliance is lowered, which is a factor that deteriorates renal function. It is known that deterioration of renal function is accompanied in 50 to 70% of patients with low bladder compliance. For patients with poor bladder compliance, a consensus has not yet been established regarding the treatment method. This is especially true in the case of drug treatment rather than surgical methods. There are limited cases where bladder compliance is improved with anticholinergics, which have been conventionally administered to the patients. According to the existing literature, increase of bladder compliance was observed in some patients with anticholinergics such as tolterodine, propiverine, and oxybutynin. But the bladder compliances were not completely normalized in every patient. Moreover, adverse effects of anticholinergics have been reported in a significant number of the patients.

The objective of this study is to analyze the effect of mirabegron (a beta3-adrenoceptor agonist) on bladder compliance in patients who had no effect on bladder compliance with prior anticholinergics treatment. In this study, low bladder compliance is defined as 20 ml/cmH2O or less.

DETAILED DESCRIPTION:
This study will be conducted as a prospective paired comparison study. In this study, low bladder compliance is defined as 20 ml/cmH2O or less. For patients who had no effect on anticholinergic treatment (at least 1 month of treatment). Mirabegron 50mg/day is administered for 8 weeks; and then, previously administered antimuscarinics were administered again for another 8 weeks. On each visit day (after 8 weeks of mirabegron, and after 8 weeks of anticholinergics), urodynamics test, voiding diary, and patient symptom questionnaire evaluations are going to be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 19 years of age
2. Bladder compliance is 20ml/cmH2O or less
3. Patient who has been treated with antimuscarinic for at least 1 month, but has not been effective.
4. Patient who agrees to and signs the informed consent

Exclusion Criteria:

1. Those who have taken clinical drugs with other ingredients (other than this experiment) for the past 60 days or participated in clinical trials using other types of medical devices.
2. Those who have previously undergone bladder augmentation
3. Those who currently have an indwelled catheter for urination
4. Those with abnormal findings in renal function (serum creatinine >2 mg/dL)
5. Those with abnormal liver function (serum AST/ALT >2 times upper limit, GGT >3 times upper limit of normal,total bilirubin >2 times upper limit of normal)
6. Those with a history of bladder cancer before screening
7. Those who were diagnosed with interstitial cystitis
8. Those with active UTI
9. Those who are pregnant or breastfeeding
10. Those with a history of previous treatment with mirabegron
11. Those who are allergic to beta 3 agonist, who are expected to be allergic to mirabegron
12. Those confirmed as resting SBP >180 mmHg and/or DBP >110 mmHg
13. Those confirmed as resting HR >100 beats per minute
14. Male patients who are likely to become pregnant or donate sperm during the study period or within 28 days of the last drug administration of the study.
15. Those who do not respond to surveys and research follow-up visits
16. Those for whom the researcher judges that the treatment method of this study is not the best treatment for the patient

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-01-12 (Actual); Primary Completion 2023-03-02 (Estimated); Study Completion 2023-03-02 (Estimated)

PRIMARY OUTCOMES:
Comparison of changes in Bladder compliance at 8 weeks after administration of each drug | Bladder compliance is assessed after 8 weeks of Mirabegron, and after 8 weeks of anticholinergics
  Bladder compliance is analyzed through urodynamic study (cystometrogram). During the cystometrogram test, the value obtained by dividing the maximum bladder volume by the detrusor pressure at end-filling is going to be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Jang Hwan Kim, Principal Investigator — Department of Urology and Urological Science Institute, Yonsei University College of Medicine, Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided